CLINICAL TRIAL: NCT06226090
Title: A Randomized, Double-blind, Placebo-controlled Phase 2 Study of TG103 Injection in the Management of Non-diabetic Overweight or Obesity
Brief Title: A Study of TG103 Injection in the Management of Non-diabetic Overweight or Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYSA1803-017
Record Dates: First submitted 2024-01-11; First posted 2024-01-26 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- TG103 7.5 mg (Experimental)
  Interventions: Drug: TG103 7.5 mg
- Placebo 7.5 mg (Placebo Comparator)
  Interventions: Drug: Placebo 7.5 mg
- TG103 15 mg (Experimental)
  Interventions: Drug: TG103 15 mg
- Placebo 15 mg (Placebo Comparator)
  Interventions: Drug: Placebo 15 mg
- TG103 22.5 mg (Experimental)
  Interventions: Drug: TG103 22.5 mg
- Placebo 22.5 mg (Placebo Comparator)
  Interventions: Drug: Placebo 22.5 mg

INTERVENTIONS:
Drug: TG103 7.5 mg — Subcutaneous injections with calorie-restricted diet and increased physical activity for 24 weeks. Dose is 7.5mg once a week.
  Arms: TG103 7.5 mg
Drug: Placebo 7.5 mg — Subcutaneous injections with calorie-restricted diet and increased physical activity for 24 weeks. Dose is 7.5mg once a week.
  Arms: Placebo 7.5 mg
Drug: TG103 15 mg — Subcutaneous injections with calorie-restricted diet and increased physical activity for 24 weeks. Doses gradually increased from 7.5 mg to 15 mg.
  Arms: TG103 15 mg
Drug: Placebo 15 mg — Subcutaneous injections with calorie-restricted diet and increased physical activity for 24 weeks. Doses gradually increased from 7.5 mg to 15 mg.
  Arms: Placebo 15 mg
Drug: TG103 22.5 mg — Subcutaneous injections with calorie-restricted diet and increased physical activity for 24 weeks. Doses gradually increased from 7.5 mg to 22.5 mg.
  Arms: TG103 22.5 mg
Drug: Placebo 22.5 mg — Subcutaneous injections with calorie-restricted diet and increased physical activity for 24 weeks. Doses gradually increased from 7.5 mg to 22.5 mg.
  Arms: Placebo 22.5 mg

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, parallel phase 2 study to evaluate efficacy, safety, pharmacokinetic characteristics and immunogenicity of TG103 injection for weight management in non-diabetic patients with overweight in the presence of comorbidities or obesity, in addition to lifestyle intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years ≤ age ≤ 75 years.
* Body Mass Index (BMI) ≥ 28 kg/m^2, or 24 kg/m^2 < BMI ≤ 28 kg/m^2 with at least one of obesity-related complications.
* Regular diet and exercise and stable body weight (i.e., self-reported body weight change < 5%) within 12 weeks before screening as well as body weight ≥ 60 kg at screening.
* Weight loss less than 5% or no weight loss after diet and exercise intervention for at least 12 weeks.

Exclusion Criteria:

* History of type 2 diabetes, type 1 diabetes or hypoglycemia.
* Overweight or obesity due to disease or drug; or weight increase due to non-fat mass increase; or monogenic obesity.
* Medications or products which are judged by investigators to cause change in weight and influence trial evaluations have been used within 12 weeks before screening or will be used during study.
* Weight loss less than 5% by monotherapy or combination with GLP-1 receptor agonists for at least 12 weeks before screening.
* Bariatric surgery within 12 months before screening; or no full recovery from any surgery or injury at screening; or gastrointestinal motility dysfunction due to gastrointestinal surgery.
* Participation in any clinical trial to receive treatment within 12 weeks before screening, or participation in clinical trial to receive TG103 before screening.
* History of allergy or suspected allergy to GLP-1 receptor agonists or antibody agents, or suspected allergy to TG103 judged by investigator due to other severe allergy history.
* Personal history or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2 (MEN-2).
* History or screening ultrasound reports of chronic pancreatitis, acute pancreatitis, etc.
* History of severe gastrointestinal disease; or gastrointestinal symptom at screening; or discontinuation of GLP-1 receptor agonist, GLP-1/GIP receptor agonist, GLP-1/GCG receptor agonist or metformin due to gastrointestinal adverse reaction.
* Severe infection at screening.
* Skin disorder that influences safety evaluation at screening.
* History of severe disease or malignant tumor.
* Systolic blood pressure ≥ 160 mmHg, diastolic blood pressure ≥ 100 mmHg, NYHA Grade Ⅲ-Ⅳ, QTc interval prolongation or severe arrhythmia at screening.
* History of abnormal thyroid function with requirement of medication treatment at screening, or screening TSH beyond the normal reference range.
* One of the followings at screening: 1) HbA1c ≥ 6.5%, or FPG ≥ 7.0mmol/L or<2.8mmol/L; 2) calcitonin ≥ 50 ng/L; 3) ALT or AST>3 × UNL (upper normal limit), or total bilirubin>1.5 × UNL; 4) blood amylase or lipase>1.5 × UNL, 5) TG>5.6mmol/L, 6) eGFR<60ml/min/1.73m^2 , 7) positive of HBsAg, HCV-antibody, HIV-antibody or anti-TP antibody, 8) WBC< 3×10^9/L, or Hb <100g/L, 9) INR>1.2.
* History of drug abuse, drug dependence or alcoholism.
* History of moderate to severe depression, or screening Patient Health Questionaire-9 (PHQ-9) score ≥ 15.
* The fertile female who is pregnant, breast-feeding or with blood HCG positive at screening; or the fertile participants and their partner cannot use an effective contraceptive method during the trial and within 3 months after the end of treatment.
* Other situations unsuitable for this study in the investigator's opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Percentage relative change from baseline in body weight at week 24 | From baseline to week 24

SECONDARY OUTCOMES:
Proportion of participants with weight loss of ≥ 5% at week 24 | From baseline to week 24
Proportion of participants with weight loss of ≥ 10% at week 24 | From baseline to week 24
Change from baseline to week 24 in waist circumference | From baseline to week 24
Relative change from baseline in body weight at week 24 | From baseline to week 24
Change from baseline to week 24 in systolic blood pressure | From baseline to week 24
Change from baseline to week 24 in diastolic blood pressure | From baseline to week 24
Title: Change from baseline to week 24 in serum total cholesterol | From baseline to week 24
Title: Change from baseline to week 24 in serum triglyceride | From baseline to week 24
Title: Change from baseline to week 24 in serum low density lipoprotein cholesterol | From baseline to week 24
Title: Change from baseline to week 24 in serum high density lipoprotein cholesterol | From baseline to week 24

OTHER OUTCOMES:
Number of TEAEs (Treatment Emergent Adverse Events) and SAEs (Serious Adverse Events) | From baseline to week 27
Change from baseline to week 24 in serum calcitonin | From baseline to week 24
Change from baseline to week 24 in serum alanine transaminase | From baseline to week 24
Change from baseline to week 24 in serum creatinine | From baseline to week 24
Change from baseline to week 24 in serum HCG (Human Chorionic Gonadotophin) | From baseline to week 24
Plasma concentration of TG103 | From baseline to week 27
Number of patients with positive TG103 antibody | From baseline to week 27

CONTACTS AND LOCATIONS:
Overall Officials: Li Yan Study Principal Investigator, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Clinical Trials Information Group, Shijiazhuang, Hebei, China